CLINICAL TRIAL: NCT06717269
Title: A Phase 1, Open-Label Study in Healthy Volunteers to Evaluate the Relative Bioavailability of NX-5948 Tablets Compared to Capsules, and the Effect of Food and an Acid-reducing Agent on the Pharmacokinetics of NX-5948
Brief Title: Relative Bioavailability of NX-5948 Tablets vs Capsules and the Effect of Covariates on the PK of NX-5948 Tablets
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NX-5948-304
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NX-5948 tablet and capsule under fasted and fed conditions (Experimental)
  Interventions: Drug: NX-5948
- NX-5948 tablet and capsule combined with esomeprazole under fasted conditions (Experimental)
  Interventions: Drug: NX-5948; Drug: Esomeprazole

INTERVENTIONS:
Drug: NX-5948 — Administered orally in tablet or capsule form
Drug: Esomeprazole — Administered orally in capsule form
  Arms: NX-5948 tablet and capsule combined with esomeprazole under fasted conditions

SUMMARY:
This is a multiple part, multiple cohort study evaluating the relative bioavailability, food effect, and drug-drug interaction of NX-5948 in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, male or female 19-55 years of age
* Continuous non-smoker who has not used nicotine and tobacco-containing products for at least 3 months prior to the first dosing
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, or 12-lead safety ECGs at the screening visit, as deemed by the PI or designee
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Key Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* Clinically significant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neoplastic myeloproliferative, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine or connective tissue diseases or disorders
* History of any gastrointestinal surgery or cholecystectomy that could impact the PK of NX-5948
* History or presence of alcohol or drug abuse within the past 2 years
* History or presence of hypersensitivity, angioedema, or idiosyncratic reaction to the study drug(s) or related compounds
* History or presence of:

  * Significant multiple and/or severe allergies, including anaphylactic reaction.
  * Personal or family history of prolonged QT syndrome or family history of sudden cardiac death.
  * Evidence of atrial fibrillation, atrial flutter, complete bundle branch block, Wolff Parkinson-White Syndrome, or cardiac pacemaker.
  * Adrenal insufficiency.
  * Skin infection.
* Female volunteers of childbearing potential
* Female volunteer with a positive pregnancy test
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit
* Donation of blood or significant blood loss within 56 days prior to the first dosing
* Plasma donation within 7 days prior to the first dosing
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* Previous exposure to NX-5948.
* Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to the first dosing, whichever is longer. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of PK parameters: NX-5948 tablets versus capsules | 9 weeks
  Relative bioavailability of NX-5948 tablet, compared to capsule, will be measured using PK parameters (AUC)
Assessment of PK parameters: NX-5948 tablets versus capsules | 9 weeks
  Relative bioavailability of NX-5948 tablet, compared to capsule, will be measured using PK parameters (Cmax)
Assessment of PK parameters NX-5948 tablets versus capsules | 9 weeks
  Relative bioavailability of NX-5948 tablet, compared to capsule, will be measured using PK parameters (Tmax)
Food effect and effect of esomeprazole on AUC0-t for single-dose NX-5948 tablet | 9 weeks
  Evaluate the effect of food and the effect of multiple doses of esomeprazole on the single-dose PK of NX-5948 tablet
Food effect and effect of esomeprazole on AUC0-inf for single-dose NX-5948 tablet | 9 weeks
  Evaluate the effect of food and the effect of multiple doses of esomeprazole on the single-dose PK of NX-5948 tablet
Food effect and effect of esomeprazole on Cmax for single-dose NX-5948 tablet | 9 weeks
  Evaluate the effect of food and the effect of multiple doses of esomeprazole on the single-dose PK of NX-5948 tablet

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nurix Therapeutics
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No